CLINICAL TRIAL: NCT05757960
Title: Effects of TMD-specific Physiotherapy in Individuals With Hypermobile Ehlers-Danlos Syndrome
Brief Title: TMD-specific Physiotherapy in hEDS Patients Individuals With Hypermobile Ehlers-Danlos Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: German Society of Craniomandibular Function and Disorders in the DGZMK. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMD_Physio_EDS
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-05

CONDITIONS: Hypermobile Ehlers-Danlos Syndrome
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3 | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physiotherapy (Experimental): Using a strictly defined physiotherapy protocol, the effects on temporomandibular dysfunctions are studied.
  Interventions: Procedure: Physiotherapy

INTERVENTIONS:
Procedure: Physiotherapy — Various physiotherapeutic techniques are used in three defined sessions. Before the first session, a dental examination is performed and a clinical functional status is obtained to assess the extent of temporomandibular dysfunction. The results are recorded on validated questionnaires.

SUMMARY:
The aim of this study is to analyze the effects of strictly defined physiotherapy in patients temporomandibular dysfunction (TMD) and hypermobile Ehlers-Danlos Syndrome (hEDS). Patients will be clinically examined before starting physiotherapy and fill in the questionnaires. Subsequently, it will be followed up whether changes occur as a result of physiotherapy.

This study is a pilot study and is intended to be hypothesis generating in nature. Based on the resulting hypothesis, it will be verified by a study with a control group.

ELIGIBILITY:
Inclusion Criteria:

1. written consent to participate in the study
2. confirmed diagnosis of hEDS (based on the diagnostic criteria of the current classification of 2017).
3. pain in the area of the masticatory muscles and/or the temporomandibular joints
4. command of the German language, both spoken and written

Exclusion Criteria:

1. currently undergoing TMD-specific treatment (physiotherapy, pain therapy masticatory muscles and/or temporomandibular joint, orthopedic treatment, osteopathic treatment).
2. persons diagnosed with depression, anxiety or stress disorder
3. taking opiates
4. pregnant women
5. minors
6. persons with mental disability
7. persons who are not able to speak and write the German language
8. persons with legal representatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of temporomandibular pain | Up to 3 months after the last physiotherapy intervention
  The German version of the Graded chronic pain scale (GCS) is used to measure the level of pain.
  The score ranges from level 0-IV, 0 representing no pain, I-II functional pain, and level III-IV dysfunctional, chronic pain.

SECONDARY OUTCOMES:
Effects on psychosocial impairment | Up to 3 months after the last physiotherapy intervention
  The German version of the Depression Anxiety Stress Scale (DASS) is used to assess psychosocial impairment.
  The scale assesses the the dimensions Depression, Anxiety and Stress. The scale comprises a total of 21 questions, 7 questions for each of the named dimensions. Each question can be answered from 0-3, 0 for no impact and 3 for highest impact. The scores for each dimension are added. An increased probability for the occurrence of depression occurs with values from 10, for anxiety from 6 and for stress from 10.
Effects on oral health-related quality of life (OHRQoL) | Up to 3 months after the last physiotherapy intervention
  The German version of the Oral Health Impact Profile (OHIP-G5) is used to assess OHRQoL. The questionnaire consists of 5 questions covering the 4 dimensions Oral Function, Orofascial Pain, Orofacial Appearance and Psychosocial impact. Each question can be answered from 0-4, where 0 stands for no impact and 4 for the highest impact. The values for the individual dimensions are formed and therefore range from 0-4 points; two questions address the Oral Function dimension, which is why values of 0-8 can be achieved here.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Oelerich, Dr. med. dent., Principal Investigator — Department for Prosthodonctics and Biomaterials, University Hospital Münster
Locations (1):
- Department for Prosthodontics and Biomaterials, University Hospital Münster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No